CLINICAL TRIAL: NCT00534092
Title: Long-term Outcomes Among Patients With Lumbar Spinal Stenosis Treated With the X STOP® Interspinous Process Decompression System: Five-Year Follow-up of IDE Patient Cohorts
Brief Title: Long-Term Outcomes for Lumbar Spinal Stenosis Patients Treated With X STOP®
Status: Completed | Type: Observational
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Other Study IDs: LSS-004-LTO
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2015-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; X STOP
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: X STOP® Interspinous Process Decompression System — The X STOP is a titanium implant that fits between the spinous processes of the lumbar spine. It is made from Ti-6AI-4V Eli titanium alloy (ISO 5832/3) and consists of two components: a spacer assembly and a wing assembly.

SUMMARY:
The Long-Term Outcomes Study (LTOS) is a multi-center longitudinal cohort study of all patients who received the X-STOP device in the Pivotal Trial, Continued Access Protocol (CAP), or Cross-over Study (COS). It is designed to supplement postmarket safety and effectiveness data to be gathered in a Condition of Approval (CoA) study of a population of patients with moderately impaired physical function who elect to undergo X-STOP surgery.

DETAILED DESCRIPTION:
Evaluate the long term safety and effectiveness of the X-Stop interspinous process decompression system In the patients who received the X-Stop under the IDE. These patients consist of two cohorts to be evaluated: patients who had moderately impaired physical function prior to X-Stop implantation (as determined by a baseline score >2.0 in the physical function (PF) domain of the Zurich claudication questionnaire), and patients who had mildly impaired physical function prior to X-Stop surgery(as determined by a baseline score <=2.0 in the PF domain of the Zurich claudication questionnaire (ZCQ), through the fifth postoperative year. Clinical examination will be performed at each office visit to confirm the absence of neurological complications. X-ray films (AP/lateral views) taken during the fifth postoperative year will, be analyzed to confirm A) maintenance of distraction and B) the absence of radiological evidence of device-related complications. Secondary endpoints will include mean scores from the SF-36, and incidence rates of adverse events, device failures, and secondary surgeries.

ELIGIBILITY:
Inclusion Criteria:

A patient will be admitted into the LTOS program if he/she meets all of the following inclusion criteria:

1. Completed participation in the Pivotal Trial, CAP, or COS and has the X STOP implant(s) intact at the time of LTOS enrollment; OR is an active CAP/COS participant, has the X STOP implant(s) intact, and has not completed a 24-month follow-up visit in his/her CAP/COS study.
2. Is willing and able to provide Informed Consent
3. Is willing and able to return to the clinic for a clinical evaluation or complete study questionnaires without a clinic visit.

Exclusion Criteria:

A patient will not be admitted into the LTOS program if he/she meets any of the following exclusion criteria:

1. Participated in the Pivotal Trial as part of the X STOP group, but the device has been removed.
2. Participated in the CAP or COS programs, but the device has been removed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received implants and completed participation in the Pivotal, CAP, or COS studies and has the implant intact and is willing and able to provide consent and return to the clinic for evaluation or complete study questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2006-12; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - St. Mary's Spine Center, San Francisco, California
  - Neurological & Spine Associates, Scarborough, Maine
  - Greater Baltimore Spine Care, Timonium, Maryland
  - Neurological Specialist, Norfolk, Virginia
  - University Hospital, Madison, Wisconsin

REFERENCES:
- [Background] Hsu KY, Zucherman JF, Hartjen CA, Mehalic TF, Implicito DA, Martin MJ, Johnson DR 2nd, Skidmore GA, Vessa PP, Dwyer JW, Cauthen JC, Ozuna RM. Quality of life of lumbar stenosis-treated patients in whom the X STOP interspinous device was implanted. J Neurosurg Spine. 2006 Dec;5(6):500-7. doi: 10.3171/spi.2006.5.6.500. PMID 17176013
- [Background] Zucherman JF, Hsu KY, Hartjen CA, Mehalic TF, Implicito DA, Martin MJ, Johnson DR 2nd, Skidmore GA, Vessa PP, Dwyer JW, Puccio ST, Cauthen JC, Ozuna RM. A multicenter, prospective, randomized trial evaluating the X STOP interspinous process decompression system for the treatment of neurogenic intermittent claudication: two-year follow-up results. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1351-8. doi: 10.1097/01.brs.0000166618.42749.d1. PMID 15959362

RESULTS

PARTICIPANT FLOW:
Groups:
- Target: Patients with impaired physical function prior to X-STOP implantation, as determined by a baseline score >2.0 in the Physical Function (PF) domain of the Zurich Claudication Questionnaire (ZCQ).
- Safety: Patients who had mildly impaired physical function prior to X-STOP implantation, as determined by a baseline score ≤2.0 in the PF domain of the ZCQ.
Period: Overall Study
Arm/Group | Target | Safety
Started | 55 | 14
Completed | 53 | 14
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — personal reasons/family concerns | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (10.2) | 76.0 (8.9) | 72.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 32 | 6 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 2
  Black or African American | 1 | 0 | 1
  Native Hawaiian / Pacific Islander | 1 | 0 | 1
  White | 46 | 12 | 58
  Unknown | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Rates (At ≥ 5 Years)
Description: Seven treatment success criteria were defined as follows: clinically significant improvement (at least 0.5 points) in Symptom Severity (SS) domain of Zurich Claudication Questionnaire (ZCQ), clinically significant improvement (at least 0.5 points) in Physical Function (PF) domain of ZCQ, Patient Satisfaction (PS) score of <2.5 points in ZCQ, no additional lumbar spinal stenosis surgery at the index level, maintenance of distraction, no device dislodgement, no device-related complications. All 7 criteria must be met to be considered a treatment success.
Time Frame: 3+ years following first 2 years post-X-STOP implant through IDE study
Population: Patients who received the X-STOP and 1) completed the IDE trial or CAP/COS under IDE #G990128 or 2) were participating in the CAP/COS program, were eligible for the LTOS study. 55 included in analysis met moderately impaired baseline physical function. 14 had mildly impaired physical function at baseline and were analyzed as separate safety cohort.
Measure: Number; unit: percentage of participants
Groups:
- Total: Total patients included target group and safety group.
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
percentage of participants
  Treatment success rate (n=49, 13, 62) | 40.8 | 30.8 | 38.7
  SS improved >=0.5 point (n=52, 13, 65) | 53.8 | 84.6 | 60.0
  PF improved >=0.5 point (n=52, 14, 66) | 73.1 | 50.0 | 68.2
  PS Score <2.5 (n=53, 14, 67) | 81.1 | 92.9 | 83.6
  No additional surgery at index level(n=53, 14, 67) | 94.3 | 100.0 | 95.5
  Maintenance of distraction (n=42, 11, 53) | 95.2 | 90.9 | 94.3
  No dislodgement of implant (n=43, 11, 54) | 100.0 | 81.8 | 96.3
  No device-related complication (n=53, 14, 67) | 94.3 | 100.0 | 92.5

2. Secondary Outcome: Change in Symptom Severity (SS) and Physical Functioning (PF) as Using Zurich Claudication Questionnaire (ZCQ) Domain Scores (At ≥ 5 Years)
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: SS, PF, and post-treatment Patient Satisfaction (PS). SS domain is based on seven questions (overall pain, pain frequency, pain in the back, pain in the leg, numbness, weakness, and balanced disturbance). The first 6 questions are scored 1 to 5. Balance disturbance is scored in a 1-3-5 scale. The SS score is the mean of all answered items in the questionnaire ranging from 1to 5. If more than two items were missing, the SS score was considered as missing. PF score is the mean of five physical function questions ranging from 1 to 4. If more than one item were missing, the PF score was considered as missing. In each domain, a lower score represents a better outcome/condition. The change is calculated as the score at 5+ years after X-STOP implantation minus the baseline score.
Time Frame: Baseline and 3+ years following first 2 years post-X-STOP implant through IDE study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
units on a scale
  Mean Change in SS (n=52, 13, 65) | -0.8 (0.9) | -1.0 (0.5) | -0.8 (0.8)
  Mean change in PF (n=52, 14, 66) | -1.0 (0.7) | -0.4 (0.4) | -0.8 (0.7)

3. Secondary Outcome: Patient Satisfaction (PS) as Assessed by Zurich Claudication Questionnaire (ZCQ) Domain Scores (At ≥ 5 Years)
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: SS, PF, and post-treatment Patient Satisfaction (PS). PS score is the mean of 6 questions scored from 1 to 4 if the number of responses exceeded four, a lower score represents a better outcome. Patients with mean scores <2.5 at 5 years postoperative evaluation were considered positive, which implied patient treatment satisfaction.
Time Frame: 3+ years following first 2 years post-X-STOP implant through IDE study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 53 | 14 | 67
units on a scale | 1.7 (0.8) | 1.5 (0.6) | 1.6 (0.7)

4. Secondary Outcome: Change in Quality of Life Using Short Form 36-Question (SF-36) Health Survey (At ≥ 5 Years)
Description: Quality of life was assessed by the SF-36 health survey. It includes 8 subdomains (bodily pain, physical functioning, role-physical, general health and vitality, social functioning, role-emotional, and mental health) and 2 component summaries (physical component summary [PCS] and mental component summary [MCS]). Scores for each subdomain and component summary range from 0 "worst" to 100 "best. The change from baseline to the 5 year postoperative visit for each of these domains is presented.
Time Frame: Baseline and 3+ years following first 2 years post-X-STOP implant through IDE study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
units on a scale
  Bodily Pain (n=52, 14, 66) | 23.4 (26.2) | 31.1 (19.9) | 25.0 (25.1)
  General Health (n=52, 14, 66) | -5.4 (14.1) | -0.9 (11.4) | -4.2 (13.6)
  MCS (n=49, 13, 62) | 3.9 (12.6) | 2.7 (8.9) | 3.7 (11.9)
  Mental Health (n=52, 14, 66) | 3.8 (19.5) | 3.4 (10.9) | 3.7 (17.9)
  PCS (n=49, 13, 62) | 8.6 (10.4) | 11.6 (9.2) | 9.2 (10.2)
  Physical Functioning (n=52, 14, 66) | 28.0 (30.0) | 27.1 (15.9) | 27.8 (27.5)
  Role-Emotional (n=50, 13, 63) | 24.0 (58.7) | 35.9 (44.0) | 26.5 (55.9)
  Role-Physical (n=50, 14, 64) | 28.5 (51.8) | 50.0 (42.7) | 33.2 (50.4)
  Social Functioning (n=52, 14, 66) | 32.0 (34.9) | 15.2 (23.1) | 28.4 (33.3)
  Vitality (n=52, 14, 66) | 7.9 (25.2) | 10.0 (14.3) | 8.3 (23.3)

5. Other Pre Specified Outcome: Number of Patients With Subsequent Lumbar Spinal Surgeries That Occurred During the Study
Description: The surgeries that occurred subsequent to the original X-STOP implantation were categorized as revision, removal, reoperation, supplemental fixation, and other.
Time Frame: 3+ years following first 2 years post-X-STOP implant through IDE study
Measure: Number; unit: participants
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
participants
  Number of Patients with Subsequent surgeries | 5 | 1 | 6
  Number of Patients with Revision | 2 | 0 | 2
  Number of Patients with Removal | 3 | 0 | 3
  Number of Patients with Re-operations | 0 | 0 | 0
  Number of Patients with Supplemental Fixations | 0 | 0 | 0
  Number of Patients with other subsequent surgeries | 2 | 1 | 3

6. Other Pre Specified Outcome: Number of Patients With Device/Procedure Related Adverse Events That Occurred During the Study
Time Frame: 3+ years following first 2 years post-X-STOP implant through IDE study
Measure: Number; unit: participants
Arm/Group | Target | Safety | Total
Number analyzed (Participants) | 55 | 14 | 69
participants
  Implant related | 0 | 0 | 0
  Procedure related | 1 | 0 | 1
  Implant & Procedure related | 2 | 0 | 2
  Undetermined | 3 | 0 | 3
  Not related | 15 | 5 | 20

ADVERSE EVENTS:
Time Frame: 3+ years following first 2 years post-X-STOP implant through IDE study
Description: An adverse event case report form was administered at each follow up visit with routine investigator assessment; adverse events were source verified.
  Patients may have had multiple adverse events.
Arm/Group | Target | Safety | Total
Serious Adverse Events (participants affected / at risk) | 11/55 | 4/14 | 15/69
Other Adverse Events (participants affected / at risk) | 48/55 | 13/14 | 61/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Target (N=55) | Safety (N=14) | Total (N=69)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Device dislocation (General disorders) | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 1
Device deployment issue (General disorders) | 1 | 0 | 1
Device failure (General disorders) | 1 | 0 | 1
Hypertrophy (General disorders) | 1 | 0 | 1
Periprosthetic fracture (General disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Spinal claudication (Nervous system disorders) | 3 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0 | 1
Hip surgery (Surgical and medical procedures) | 1 | 0 | 1
Intervertebral disc operation (Surgical and medical procedures) | 0 | 1 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Target (N=55) | Safety (N=14) | Total (N=69)
arrhythmia (Cardiac disorders) | 0 | 1 | 1
atrial fibrillation (Cardiac disorders) | 2 | 1 | 3
coronary artery disease (Cardiac disorders) | 1 | 0 | 1
myocardial infarction (Cardiac disorders) | 2 | 0 | 2
factor v leiden mutation (Congenital, familial and genetic disorders) | 1 | 0 | 1
deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 1
hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 1
acromegaly (Endocrine disorders) | 1 | 0 | 1
thyroid disorder (Endocrine disorders) | 1 | 0 | 1
cataract (Eye disorders) | 1 | 1 | 2
glaucoma (Eye disorders) | 2 | 1 | 3
macular degeneration (Eye disorders) | 1 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1 | 1
dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 4 | 6
haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2
nausea (Gastrointestinal disorders) | 1 | 0 | 1
oesophageal stenosis (Gastrointestinal disorders) | 2 | 0 | 2
vomiting (Gastrointestinal disorders) | 1 | 0 | 1
asthenia (General disorders) | 1 | 0 | 1
chills (General disorders) | 1 | 0 | 1
drug withdrawal syndrome (General disorders) | 0 | 1 | 1
fatigue (General disorders) | 1 | 0 | 1
feeling abnormal (General disorders) | 0 | 1 | 1
hernia (General disorders) | 1 | 0 | 1
oedema peripheral (General disorders) | 1 | 0 | 1
pain (General disorders) | 0 | 1 | 1
polyp (General disorders) | 1 | 0 | 1
multiple allergies (Immune system disorders) | 0 | 3 | 3
bronchitis (Infections and infestations) | 0 | 1 | 1
cellulitis (Infections and infestations) | 1 | 0 | 1
cystitis (Infections and infestations) | 1 | 1 | 2
influenza (Infections and infestations) | 1 | 0 | 1
pneumonia (Infections and infestations) | 1 | 1 | 2
upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
urinary tract infection (Infections and infestations) | 2 | 0 | 2
ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
fall (Injury, poisoning and procedural complications) | 6 | 0 | 6
femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
road traffic accident (Injury, poisoning and procedural complications) | 3 | 1 | 4
spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
pedal pulse decreased (Investigations) | 1 | 0 | 1
diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 3
gout (Metabolism and nutrition disorders) | 0 | 2 | 2
hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
hypocholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0 | 9
arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6
arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 13 | 2 | 15
bursitis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5
polychondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
malignant neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3
amnesia (Nervous system disorders) | 1 | 0 | 1
ataxia (Nervous system disorders) | 1 | 0 | 1
carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
carpal tunnel syndrome (Nervous system disorders) | 2 | 0 | 2
cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
cognitive disorder (Nervous system disorders) | 1 | 1 | 2
cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
headache (Nervous system disorders) | 1 | 1 | 2
hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
occipital neuralgia (Nervous system disorders) | 1 | 0 | 1
parkinson's disease (Nervous system disorders) | 1 | 0 | 1
peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 1
radicular pain (Nervous system disorders) | 2 | 1 | 3
sciatica (Nervous system disorders) | 2 | 0 | 2
spinal claudication (Nervous system disorders) | 4 | 0 | 4
transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
vascular dementia (Nervous system disorders) | 1 | 0 | 1
anxiety (Psychiatric disorders) | 1 | 0 | 1
depression (Psychiatric disorders) | 2 | 1 | 3
depressive symptom (Psychiatric disorders) | 1 | 0 | 1
insomnia (Psychiatric disorders) | 0 | 1 | 1
incontinence (Renal and urinary disorders) | 1 | 0 | 1
pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
proteinuria (Renal and urinary disorders) | 1 | 0 | 1
benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2 | 4
prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 1
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
bladder repair (Surgical and medical procedures) | 0 | 2 | 2
cholecystectomy (Surgical and medical procedures) | 1 | 1 | 2
corneal transplant (Surgical and medical procedures) | 1 | 0 | 1
hip arthroplasty (Surgical and medical procedures) | 2 | 1 | 3
injection (Surgical and medical procedures) | 1 | 0 | 1
knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
knee operation (Surgical and medical procedures) | 1 | 0 | 1
partial lung resection (Surgical and medical procedures) | 1 | 0 | 1
spinal operation (Surgical and medical procedures) | 1 | 0 | 1
stent placement (Surgical and medical procedures) | 2 | 0 | 2
wound treatment (Surgical and medical procedures) | 0 | 1 | 1
aortic aneurysm (Vascular disorders) | 1 | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
hot flush (Vascular disorders) | 1 | 0 | 1
hypertension (Vascular disorders) | 6 | 1 | 7
intermittent claudication (Vascular disorders) | 1 | 0 | 1
peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 1
phlebitis (Vascular disorders) | 1 | 0 | 1
varicose vein (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other